CLINICAL TRIAL: NCT07323589
Title: Impact of Myo-Inositol vs Combined Myo-Inositol and Metformin Therapy on Conception Rates, Treatment Adherence, and Tolerability in Overweight Women Diagnosed With PCOS: A Randomized Controlled Study
Brief Title: Impact of Myo-Inositol Alone vs Myo-Inositol Plus Metformin on Conception, Adherence, and Tolerability in PCOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PAEC general hospital (Other Government)
Responsible Party: Principal Investigator, Maria Amin, Postgraduate Resident Gynecology and Obstetrics, PAEC general hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGHI-IRB(DME)-RCD-06-097
Record Dates: First submitted 2025-11-14; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: Myo-inositol; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol; Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- arm 1 (Experimental): in the comparison group of study: Researchers will compare Group A (myo-inositol 4 g/day)
  Interventions: Drug: Myoinositol
- arm 2 (Experimental): group B will be a combination group (Metformin 1500mg per day and Myo inositol 4gram per day)
  Interventions: Drug: Myoinositol; Drug: Metformin 1500 mg daily

INTERVENTIONS:
Drug: Myoinositol — myo-inositol (4 g/day)
Drug: Metformin 1500 mg daily — metfromin plus myoinositol 1500mg and 4gram per day respectively
  Arms: arm 2

SUMMARY:
The goal of this clinical trial (prospective randomized controlled trial) is to compare whether myo-inositol alone or in combination with metformin can improve conception rates, treatment compliance, and side-effect profiles in overweight women (BMI ≥25 kg/m²) diagnosed with polycystic ovary syndrome (PCOS).

The main questions it aims to answer are:

1. Does myo-inositol alone achieve conception rates comparable to the combination of myo-inositol and metformin?
2. Does the combination therapy result in more side effects and lower compliance compared to myo-inositol alone? If there is a comparison group: Researchers will compare Group A (myo-inositol 4 g/day) with Group B (myo-inositol 4 g/day + metformin 1500 mg/day) to see if the addition of metformin improves conception outcomes but at the cost of tolerability.

Participants will:

* Be randomly assigned to receive either myo-inositol alone or myo-inositol plus metformin for six months.
* Attend follow-up visits for monitoring of pregnancy outcomes confirmed by ultrasound.
* Report any side effects experienced during treatment.
* Provide information on treatment adherence and dropout rates.
* Be assessed for menstrual regularity and ovulation rates.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 35 years
* BMI ≥25 kg/m²
* Fulfilled at least two of the three Rotterdam criteria for PCOS
* Attempting to conceive naturally
* No use of hormonal drugs or insulin-sensitizers in the past three months

Exclusion Criteria:

* Endocrine disorders (e.g., diabetes, thyroid dysfunction)
* Hepatic impairment
* Kidney disease
* Gastrointestinal or malabsorption issues (IBS, IBD, celiac disease)
* Known allergies to metformin or inositol
* Pregnant or breastfeeding

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females of reproductive age group
Enrollment: 120 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Confirmed Clinical Pregnancy by Ultrasound | Up to 6 months or until pregnancy is confirmed
  Clinical pregnancy defined as the presence of a gestational sac confirmed by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Amin, Principal Investigator — PAEC general hospital, H-11/4, islamabad
Locations (1):
- PAEC general hospital, Islamabad, Isb, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agrawal A, Mahey R, Kachhawa G, Khadgawat R, Vanamail P, Kriplani A. Comparison of metformin plus myoinositol vs metformin alone in PCOS women undergoing ovulation induction cycles: randomized controlled trial. Gynecol Endocrinol. 2019 Jun;35(6):511-514. doi: 10.1080/09513590.2018.1549656. Epub 2019 Jan 7. PMID 30614289
- [Result] Thakur SS, Anjum S, Siddiqui SS. Randomised controlled trial: comparing effects of metformin versus myoinositol versus metformin and myoinositol on ovarian functions and metabolic factors in polycystic ovarian syndrome. Int J Reprod Contracept Obstet Gynecol. 2020;9(6):2542 50. doi:10.18203/2320-1770.ijrcog20202030

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-12-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT07323589/Prot_ICF_000.pdf